CLINICAL TRIAL: NCT02146625
Title: A Dose-block Randomized, Single-blind, Placebo-controlled, Single-dosing, Dose-escalation Phase I Clinical Trial to Investigate the Safety/Tolerability and Pharmacokinetics/Pharmacodynamics of CJ-40002 After Subcutaneous Injection in Healthy Adult Male Volunteers
Brief Title: Safety, Tolerability, PK, PD, ADA of Escalating Single Dose of CJ-40002 in Healthy Male Subjects
Acronym: hGH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CJ_HGH_101
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose level 1 of CJ-40002 (Experimental): * Single dose
  * 8 volunteers will be administered dose level 1 of CJ-40002 or placebo comparators.(CJ-40002:placebo=6:2)
  Interventions: Drug: CJ-40002
- Dose level 2 of CJ-40002 (Experimental): * Single dose
  * 8 volunteers will be administered dose level 2 of CJ-40002 or placebo comparators.(CJ-40002:placebo=6:2)
  Interventions: Drug: CJ-40002
- Dose level 3 of CJ-40002 (Experimental): * Single dose
  * 8 volunteers will be administered dose level 3 of CJ-40002 or placebo comparators.(CJ-40002:placebo=6:2)
  Interventions: Drug: CJ-40002
- Dose level 4 of CJ-40002 (Experimental): * Single dose
  * 8 volunteers will be administered dose level 4 of CJ-40002 or placebo comparators.(CJ-40002:placebo=6:2)
  Interventions: Drug: CJ-40002
- Dose level 5 of CJ-40002 (Experimental): * Single dose
  * 8 volunteers will be administered dose level 5 of CJ-40002 or placebo comparators.(CJ-40002:placebo=6:2)
  Interventions: Drug: CJ-40002

INTERVENTIONS:
Drug: CJ-40002

SUMMARY:
The objectives of this study are:

* To evaluate the safety and tolerability of CJ-40002 after single SC injection in healthy male volunteers.
* To evaluate the PK of CJ-40002 after single SC injection in healthy male volunteers.
* To evaluate the PD of CJ-40002 after single SC injection in healthy male volunteers.
* To evaluate the ADA of CJ-40002 after single SC injection in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers in the age between 19 and 45 years old (inclusive)
* Body mass index (BMI) in the range of 18.5 to 25 kg/m2 and weighing at least 55 kg
* Subject who have voluntarily agreed to participate in the trial and signed the written informed consent form, after having listened to the purpose, method, and effect of the clinical trial

Exclusion Criteria:

* History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, musculoskeletal or cardiovascular disease or any other condition
* History of allergy or sensitivity to any drug
* Subject with the following clinically significant laboratory abnormalities:

  * AST or ALT > 1.25 x Upper Limit Normal (ULN)
  * Total bilirubin > 1.5 x Upper Limit Normal (ULN)
  * CPK > 1.5 x Upper Limit Normal (ULN)
  * eGFR < 60 mL/min/1.73 m2
* Systolic blood pressure outside the range of 90 to 150 mmHg or diastolic blood pressure outside the range of 50 to 100 mmHg
* History of drug abuse
* History of caffeine, alcohol, smoking abuse
* Participation in any clinical investigation within 60days prior to study medication dosing
* Subjects with whole blood donation within 60days, component blood donation within 30days prior to study medication dosing
* Positive test results for HBs Ab, HCV Ab, HIV test
* Subjects considered as unsuitable based on medical judgement by investigators

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: AUC, Cmax | 15 days
Safety and Tolerability (AE's, vital signs, ECG, laboratory tests, local reaction) | 29 days

SECONDARY OUTCOMES:
Pharmacokinetics: Tmax, T1/2, CL/F, Vd | 15 days
Pharmacodynamics: Serum IGF-1, free IGF-1, IGFBP-3, GHBP | 15 days
Formation of anti-drug antibodies | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, MD, PhD, Principal Investigator — Yonsei University College of Medicine, Seoul, Korea